CLINICAL TRIAL: NCT04597190
Title: Comparative Effectiveness PTSD Trial of Sequenced Pharmacotherapy and Psychotherapy in Primary Care
Brief Title: Sequenced Treatment Effectiveness for Posttraumatic Stress
Acronym: STEPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Stanford University (Other); Boston University (Other); Washington State University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, John Cooper Fortney, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00011185
Record Dates: First submitted 2020-10-01; First posted 2020-10-22 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: PTSD
Keywords: antidepressants; exposure therapy; primary care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to treatment sequences, stratified by site and baseline antidepressant use.
Who Masked: Outcomes Assessor
Masking Description: The survey team members will be masked to which arm the study participant has been randomized.
  The PI, Co-PIs, and Co-Is will not have access to the outcomes until the primary data collection phase has been completed. The statistician will present outcomes by arm to the Data Safety Monitoring Board (DSMB) members during closed sessions of DSMB meetings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SSRI Then Augmentation by WET (Active Comparator): Prescribers will prescribe one of three SSRIs (sertraline, fluoxetine or paroxetine). Patients who do not respond to treatment by four months will have their treatment augmented by Written Exposure Therapy (WET) delivered by an integrated behavioral health consultant.
  Interventions: Drug: Selective serotonin reuptake inhibitor; Behavioral: Written Exposure Therapy
- SSRI Then Switch to SNRI (Active Comparator): Prescribers will prescribe one of three SSRIs (sertraline, fluoxetine or paroxetine). Patients who do not respond to treatment by four months will have their treatment switched to the SNRI (serotonin-norepinephrine reuptake Inhibitor) venlafaxine.
  Interventions: Drug: Selective serotonin reuptake inhibitor; Drug: Serotonin-norepinephrine reuptake inhibitor
- WET Then Switch to SSRI (Active Comparator): Integrated behavioral health consultants will deliver WET. Patients who do not respond to treatment by four months will be switched to one of three SSRIs (sertraline, fluoxetine or paroxetine).
  Interventions: Drug: Selective serotonin reuptake inhibitor; Behavioral: Written Exposure Therapy

INTERVENTIONS:
Drug: Selective serotonin reuptake inhibitor — Prescribers and patients choose among three selective serotonin reuptake inhibitors (SSRI), sertraline, paroxetine, or fluoxetine based on patient's treatment history (i.e., failed SSRI trials due to side-effects or lack of efficacy) and preference. If a patient experiences problematic side effects after taking their choice of SSRI, the provider may switch them to another of the SSRI options during the first 8 weeks of follow-up. Patients on any antidepressant (including SSRIs) at enrollment will be cross-tapered over four weeks to either fluoxetine, sertraline or paroxetine (i.e., the old drug will be tapered down while the new drug is tapering up).
Drug: Serotonin-norepinephrine reuptake inhibitor — Prescribers will prescribe venlafaxine.
  Arms: SSRI Then Switch to SNRI
Behavioral: Written Exposure Therapy — Written Exposure Therapy will be delivered during six 30 minute sessions. The first session includes psychoeducation about symptoms of PTSD, provides a treatment rationale for approaching the trauma memory, and discusses the use of writing as a means of doing so. In sessions 2-6, patients will write about the memory of their worst traumatic event for 20 minutes, with a focus on details of the event and thoughts and feelings that occurred during the event. Patients are directed to write about the same trauma memory during each session. The session ends with the therapist instructing the patient to allow themselves to experience any trauma-related memories, images, thoughts, and feelings in the interval between sessions. The therapist reads the narrative between sessions to make sure instructions were followed. Feedback about the narrative is provided to the patient at the beginning of sessions 3-6. This feedback is used to prompt the patient for writing in the current session.
  Arms: SSRI Then Augmentation by WET; WET Then Switch to SSRI

SUMMARY:
Individuals with PTSD are more likely to engage in unhealthy behaviors such as tobacco use, drug use, alcohol misuse, and have high rates of morbidity/mortality. PTSD negatively impacts marriages, educational attainment, and occupational functioning. Some patients with PTSD can be successfully referred to specialty mental health clinics, but most patients with PTSD cannot engage in specialty care because of geographical, financial and cultural barriers and must be treated in primary care. However, policy makers do not know the best way to treat PTSD in primary care clinics, especially for patients who do not respond to the initial treatment choice. There are effective treatments for PTSD that are feasible to deliver in primary care. These treatments include commonly prescribed antidepressants and brief exposure-based therapies. However, because there are no head-to-head comparisons between pharmacotherapy and psychotherapy in primary care settings, primary care providers do not know which treatments to recommend to their patients. In addition, despite high treatment non-response rates, very few studies have examined which treatment should be recommend next when patients do not respond well to the first, and no such studies have been conducted in primary care settings.

This trial will be conducted in Federally Qualified Health Centers and VA Medical Centers, where the prevalence of both past trauma exposure and PTSD are particularly high. The investigators will enroll 700 primary care patients. The investigators propose to 1) compare outcomes among patients randomized to initially receive pharmacotherapy or brief psychotherapy, 2) compare outcomes among patients randomized to treatment sequences (i.e., switching and augmenting) for patients not responding to the initial treatment and 3) examine variation in treatment outcomes among different subgroups of patients. Telephone and web surveys will be used to assessed outcomes important to patients, like self-reported symptom burden, side-effects, health related quality of life, and recovery outcomes, at baseline, 4 and 8 months. Results will help patients and primary care providers choose which treatment to try first and which treatment to try second if the first is not effective.

DETAILED DESCRIPTION:
Background: In primary care settings, PTSD frequently goes undetected and untreated. When PTSD is diagnosed in primary care, treatment is usually inadequate and outcomes are poor. This is highly problematic because many patients with PTSD prefer receiving care in primary care settings, and less than half are successfully referred to the specialty mental health setting. This is especially a concern for safety net primary settings such as Federally Qualified Health Centers and VA Medical Centers, where the prevalence of both past trauma exposure and PTSD are particularly high. However, there are effective pharmacotherapy and psychotherapy treatments for PTSD that are feasible to deliver in primary care.

Objective: Because there are no head-to-head comparisons of pharmacotherapy and psychotherapy for PTSD among primary care patients, the investigators propose to 1) compare outcomes among patients randomized to initially receive pharmacotherapy or brief psychotherapy, 2) compare outcomes among patients randomized to treatment sequences (i.e., switching and augmenting) for patients not responding to the initial treatment and 3) examine variation in treatment outcomes among different subgroups of patients.

Methods: This multi-site trial will enroll 700 patients meeting clinical criteria for PTSD from 7 Federally Qualified Health Centers and 8 VA Medical Centers. The pharmacotherapy treatments are sertraline, fluoxetine, paroxetine and venlafaxine. The psychotherapy treatment is Written Exposure Therapy. Telephone and web surveys will be used to assessed outcomes (patient treatment engagement, self-reported symptom burden, health related quality of life, and recovery outcomes) at baseline, 4 and 8 months. Patients will be the unit of the intent-to-treat analysis. Multiple imputation will be used for missing data. Mixed-models will be used to test hypotheses.

Significance: Due to a lack of head-to-head comparisons between pharmacotherapy and psychotherapy protocols, clinical practice guidelines for PTSD provide contradictory recommendations about pharmacotherapy and psychotherapy. In particular, PTSD clinical practice guidelines have little to offer primary care providers because so few trials have been conducted in this setting. The proposed large pragmatic trial will compare, head-to-head, FDA approved PTSD medications with a brief trauma-focused psychotherapy that is evidence-based and feasible to deliver in primary care. In addition, despite high treatment non-response rates, very few trials have examined treatment sequencing and none have done so in the primary care setting. For patients not responding to the initial treatment, the proposed research is powered to compare, head-to-head, alternative treatment sequences that are feasible to deliver in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Screen positive for PTSD (PC-PTSD>=3 AND PCL>=33)
* Screen positive for trauma (Brief Trauma questionnaire)

Exclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder or dementia
* Current prescription of venlafaxine
* Change in any psychotropic prescription in the past 2 months
* A scheduled specialty mental health appointment or preference for specialty mental health care
* Pregnant
* Terminally ill
* Prisoner
* Unable to communicate in English or Spanish
* <18 years of age
* Impaired decision making capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Little Rock VA Medical Center, North Little Rock, Arkansas
  - East Arkansas Family Health Center, West Memphis, Arkansas
  - Neighborhood Healthcare, San Diego, California
  - San Diego VA Medical Center, San Diego, California
  - VA Eastern Colorado Health Care, Aurora, Colorado
  - Bedford VA Medical Center, Bedford, Massachusetts
  - Ann Arbor VA Medical Center, Ann Arbor, Michigan
  - Upper Great Lakes Family Health Center, Hancock, Michigan
  - Family Medical Center of Michigan, Temperance, Michigan
  - Partnership Health Center, Missoula, Montana
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Portland VA Medical Center, Portland, Oregon
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - North Central Texas Community Health Center, Wichita Falls, Texas
  - Healthpoint, SeaTac, Washington

IPD SHARING:
Plan to Share IPD: Yes
A public use dataset will be hosted by the Patient-Centered Outcomes Research Institute Data Repository hosted by Inter-university Consortium for Political and Social Research (ICPSR), the University of Michigan's Institute for Social Research.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Fortney JC, Kaysen DL, Engel CC, Cerimele JM, Nolan JP Jr, Chase E, Blanchard BE, Hauge S, Bechtel J, Taylor A, Acierno R, Nagel N, Sripada RK, Painter JT, DeBeer BB, Zimberoff A, Bluett EJ, Teo AR, Morland LA, Grubbs K, Sloan DM, Marx BP, Heagerty PJ. Pragmatic Comparative Effectiveness of Primary Care Treatments for Posttraumatic Stress Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Dec 1;82(12):1203-1215. doi: 10.1001/jamapsychiatry.2025.2962. PMID 41091477

RESULTS

PARTICIPANT FLOW:
Groups:
- SSRI Then Augmentation by WET: Prescribers will prescribe one of three SSRIs (sertraline, fluoxetine or paroxetine). Patients who do not respond to treatment by four months will have their treatment augmented by Written Exposure Therapy (WET) delivered by an integrated behavioral health consultant.
  Selective serotonin reuptake inhibitor: Prescribers and patients choose among three selective serotonin reuptake inhibitors (SSRI), sertraline, paroxetine, or fluoxetine. If a patient experiences problematic side effects after taking their choice of SSRI, the provider may switch them to another of the SSRI options during the first 8 weeks of follow-up. Patients on any antidepressant (including SSRIs) at enrollment will be cross-tapered over four weeks to either fluoxetine, sertraline or paroxetine.
  Written Exposure Therapy: Written Exposure Therapy will be delivered during six 30 minute sessions. The first session includes psychoeducation. In sessions 2-6, patients will write about the memory of their worst traumatic event for 20 minutes, with a focus on details of the event and thoughts and feelings that occurred during the event. Patients are directed to write about the same trauma memory during each session. The therapist reads the narrative between sessions to make sure instructions were followed. Feedback about the narrative is provided to the patient at the beginning of sessions 3-6. This feedback is used to prompt the patient for writing in the current session.
- WET Then Switch to SSRI: Integrated behavioral health consultants will deliver WET. Patients who do not respond to treatment by four months will be switched to one of three SSRIs (sertraline, fluoxetine or paroxetine).
  Written Exposure Therapy: Written Exposure Therapy will be delivered during six 30 minute sessions. The first session includes psychoeducation. In sessions 2-6, patients will write about the memory of their worst traumatic event for 20 minutes, with a focus on details of the event and thoughts and feelings that occurred during the event. Patients are directed to write about the same trauma memory during each session. The therapist reads the narrative between sessions to make sure instructions were followed. Feedback about the narrative is provided to the patient at the beginning of sessions 3-6. This feedback is used to prompt the patient for writing in the current session.
  Selective serotonin reuptake inhibitor: Prescribers and patients choose among three selective serotonin reuptake inhibitors (SSRI), sertraline, paroxetine, or fluoxetine. If a patient experiences problematic side effects after taking their choice of SSRI, the provider may switch them to another of the SSRI options during the first 8 weeks of follow-up. Patients on any antidepressant (including SSRIs) at enrollment will be cross-tapered over four weeks to either fluoxetine, sertraline or paroxetine.
Period: Overall Study
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
Started | 169 | 179 | 352
Completed | 145 | 150 | 295
Not Completed | 24 | 29 | 57

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI | Total
Number analyzed (Participants) | 169 | 179 | 352 | 700
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (15.1) | 44.4 (15.6) | 44.8 (15.4) | 45.1 (15.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 98 | 93 | 177 | 368
  Woman | 44 | 49 | 119 | 212
  Transgender Man | 0 | 1 | 0 | 1
  Transgender Women | 0 | 1 | 0 | 1
  Non-binary or gender fluid | 1 | 3 | 3 | 7
  Another identity | 1 | 1 | 2 | 4
  Missing | 25 | 31 | 51 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 28 | 51 | 100
  Not Hispanic or Latino | 110 | 105 | 222 | 437
  Unknown or Not Reported | 38 | 46 | 79 | 163
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian, Alaskan Native, or other Indigenous group | 0 | 5 | 3 | 8
  Arab or Middle Eastern | 3 | 1 | 0 | 4
  Asian | 2 | 8 | 12 | 22
  Black or African American | 30 | 28 | 70 | 128
  Multi-race | 11 | 10 | 27 | 48
  Native Hawaiian or Pacific Islander | 1 | 1 | 4 | 6
  White | 92 | 94 | 183 | 369
  Another Identity | 4 | 8 | 11 | 23
  Missing | 26 | 24 | 42 | 92
Region of Enrollment [Number; unit: participants]
  United States | 169 | 179 | 352 | 700
PTSD Check List (PCL-5) [Mean (Standard Deviation); unit: units on a scale (range 0-80)] — 20-item measure of PTSD symptom severity (range 0-80). Higher scores represent greater severity. Cutoff score of 33 is considered a positive screen for PTSD.
  units on a scale (range 0-80) | 53.2 (11.5) | 52.8 (10.9) | 52.6 (11.0) | 52.8 (11.1)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptoms
Description: Self reported burden of PTSD symptoms (PCL-5) (range 0-80, higher scores are worse)
Time Frame: 4 months (Hypothesis 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
Number analyzed (Participants) | 145 | 150 | 295
units on a scale | 39.3 (17.8) | 38.6 (17.0) | 40.5 (18.4)

2. Primary Outcome: PTSD Symptoms
Description: Self reported burden of PTSD symptoms (PCL-5) (range 0-80, higher scores are worse)
Time Frame: 8 Months (Hypotheses 2a and 2b)
Population: Participants not responding to treatment at 4-months who completed the 8-month survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
Number analyzed (Participants) | 52 | 54 | 124
units on a scale | 49.3 (17.0) | 42.1 (17.2) | 44.5 (17.3)

3. Secondary Outcome: Mental Health Related Quality of Life: SF-12V, Mental Health Component Summary Score
Description: SF-12V, Mental Health Component Summary Score (range 0-100, higher scores are better)
Time Frame: 4 months (Hypothesis 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
Number analyzed (Participants) | 145 | 150 | 293
units on a scale | 34.7 (11.6) | 34.1 (12.2) | 32.9 (11.0)

4. Secondary Outcome: Mental Health Related Quality of Life: SF-12V, Mental Health Component Summary Score
Description: SF-12V, Mental Health Component Summary Score (range 0-100, higher scores are better)
Time Frame: 8 Months (Hypotheses 2a and 2b)
Population: Participants not responding to treatment at 4-months who completed the 8-month survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
Number analyzed (Participants) | 52 | 54 | 124
units on a scale | 29.4 (12.3) | 32.0 (12.8) | 31.7 (12.2)

5. Secondary Outcome: Depression Symptoms
Description: Self reported burden of depression symptoms (PHQ-9) (range 0-27, higher scores are worse)
Time Frame: 4 months (Hypothesis 1)
Population: Participants completing the 4-month survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
Number analyzed (Participants) | 141 | 156 | 314
units on a scale | 12.6 (6.0) | 12.3 (5.9) | 13.3 (6.2)

6. Secondary Outcome: Depression Symptoms
Description: Self reported burden of depression symptoms (PHQ-9) (range 0-27, higher scores are worse)
Time Frame: 8 Months (Hypotheses 2a and 2b)
Population: Participants not responding to treatment at 4-months who completed the 8-month survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
Number analyzed (Participants) | 52 | 54 | 124
units on a scale | 14.3 (6.4) | 13.4 (5.7) | 14.6 (6.1)

7. Secondary Outcome: Generalized Anxiety Symptoms
Description: Self reported burden of anxiety symptoms (GAD-7) (range 0-21, higher scores are worse)
Time Frame: 4 months (Hypothesis 1)
Population: Participants completing the survey at 4-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
Number analyzed (Participants) | 144 | 149 | 290
units on a scale | 10.7 (5.5) | 10.4 (5.2) | 11.2 (6.0)

8. Secondary Outcome: Generalized Anxiety Symptoms
Description: Self reported burden of anxiety symptoms (GAD-7) (range 0-21, higher scores are worse)
Time Frame: 8 Months (Hypotheses 2a and 2b)
Population: Participants not responding to treatment at 4-months who completed the 8-month survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
Number analyzed (Participants) | 52 | 54 | 121
units on a scale | 12.5 (5.5) | 11.8 (5.7) | 12.9 (5.6)

9. Other Pre Specified Outcome: Number of Severe and Moderate Side Effects
Description: Self reported severity of specific side-effects
Time Frame: 4 months (Hypothesis 1)
Population: Participants completing the 4-month survey
Measure: Mean (Standard Deviation); unit: Number of side-effects
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
Number analyzed (Participants) | 53 | 54 | 126
Number of side-effects | 2.9 (2.7) | 2.6 (2.5) | 2.9 (2.4)

10. Other Pre Specified Outcome: Number of Severe and Moderate Side Effects
Description: Self reported severity of specific side-effects
Time Frame: 8 Months (Hypotheses 2a and 2b)
Population: Participants not responding to treatment at 4-months who completed the 8-month survey
Measure: Mean (Standard Deviation); unit: Number of side-effects
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
Number analyzed (Participants) | 53 | 54 | 126
Number of side-effects | 3.3 (2.2) | 2.9 (2.6) | 3.2 (2.6)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | SSRI Then Augmentation by WET | SSRI Then Switch to SNRI | WET Then Switch to SSRI
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/179 | 1/352
Serious Adverse Events (participants affected / at risk) | 32/169 | 34/179 | 63/352
Other Adverse Events (participants affected / at risk) | 34/169 | 35/179 | 60/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSRI Then Augmentation by WET (N=169) | SSRI Then Switch to SNRI (N=179) | WET Then Switch to SSRI (N=352)
Hospitalization (Investigations) | 1 (1) | 3 (3) | 7 (7)
Emergency Department Admission (Investigations) | 0 (0) | 1 (1) | 9 (9)
Suicide Intent (Investigations) | 31 (31) | 30 (30) | 46 (46)
Other (Investigations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSRI Then Augmentation by WET (N=169) | SSRI Then Switch to SNRI (N=179) | WET Then Switch to SSRI (N=352)
Increase in suicide ideation (Investigations) | 33 (33) | 35 (35) | 60 (60)
Non-suicidal injury (Investigations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT04597190/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT04597190/SAP_001.pdf